CLINICAL TRIAL: NCT02336438
Title: The Effect of Glucomannan Soluble Fiber on Glucose Homeostasis in Patients With RNY Gastric Bypass Surgery
Brief Title: The Effect of Glucomannan Soluble Fiber on Glucose Homeostasis in Patients With Roux En Y (RNY) Gastric Bypass Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bassett Healthcare (Other)
Responsible Party: Principal Investigator, Amy Freeth, Attending Physician - Endocrinology, Bassett Healthcare
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1036
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Results first posted 2015-09-21 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-01

CONDITIONS: Hypoglycemia
MeSH Terms: conditions — Hypoglycemia | interventions — (1-6)-alpha-glucomannan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baseline Phase (Control) (No Intervention): iPro CGM device will be worn for next 5 days. The subjects will maintain a diet history and will be given a One Touch glucometer and strips to check their blood glucose at home four times a day for next five days and log this onto the System Patient Log (included).
  Subjects will undergo MMTT, which includes consumption of a standard meal (Boost) and scheduled blood draws over 3 hours.
- Treatment Phase (Glucomannan) (Experimental): iPro CGM device will be worn for next 5 days. The subjects will maintain a diet history and will be given a One Touch glucometer and strips to check their blood glucose at home four times a day for next five days and log this onto the System Patient Log (included).
  Subjects will undergo MMTT, which includes consumption of a standard meal (Boost) + 5 grams of Glucomannan soluble fiber powder and scheduled blood draws over 3 hours.
  For the next five days subjects will take the following amounts of Glucomannan soluble fiber (provided by the investigator) three times a day with meals.
  Interventions: Dietary Supplement: glucomannan

INTERVENTIONS:
Dietary Supplement: glucomannan — Glucomannan is a natural, odorless soluble fiber that is found in the konjac plant. It will be given during the Intervention Phase in conjunction with the MMTT and then for 5 days at home with meals.
  Arms: Treatment Phase (Glucomannan)

SUMMARY:
One of the emerging complications of RNY gastric bypass surgery is mild to severe refractory/ recurrent postprandial hypoglycemia. This complication can lead to a significant reduction in quality of life to severe disability. Unfortunately at this time there are no treatment guidelines or proven therapeutic options for the treatment of this complication. One of the proposed treatment options is the use of fiber supplements to help modify the absorption of glucose, slow the food bolus transit time more toward normal and restore the postprandial (after meal) glucose homeostasis. The investigators are proposing a pilot project for the use of Glucomannan soluble fiber as a treatment option for postprandial hypoglycemia in this cohort. This project will help the investigators to identify if Glucomannan soluble fiber can be used as an effective dietary supplement to eliminate or reduce this condition

DETAILED DESCRIPTION:
Currently there are no therapeutic guidelines and no proven therapy available to reduce hypoglycemic episodes post RNY gastric bypass. A study done in 1988 (n=8/ patients with partial gastrectomy and hypoglycemia) showed improvement in plasma glucose level and peak insulin response in patients suffering from this complication and who were given Glucomannan soluble fiber with a standard meal. Glucomannan is a natural, odorless soluble fiber that is found in the konjac plant. The konjac glucomannan is the most viscosity food gum in nature. It has about ten times the viscosity than the cornstarch. Unfortunately no further studies have been done so far to validate or support this therapy in patients with RNY gastric bypass. This study will be the first one to see effectiveness of Glucomannan, exclusively in patients who are post RNY gastric bypass and have a diagnosis of postprandial hypoglycemia.

Visit 1: consent and screening bloodwork: Thyroid Stimulating Hormone (TSH), Free T4, Cortisol, Creatinine, and Insulin-like Growth Factor (IGF)

Visit 2: iPro Continuous glucose monitor (CGM) device will be placed and will be worn for next 5 days. The subjects will maintain a diet history and will be given a One Touch glucometer and strips to check their blood glucose at home four times a day for next five days and log this onto the System Patient Log (included).

Subjects will undergo a mixed meal tolerance test (MMTT), a, which includes consumption of a after a standard meal (Boost) and scheduled blood draws over 3 hours.

Visit 3: The subject will return to the research coordinator for the iPRO® Continuous Glucose Monitor (CGM) removal and data download from the device. After physical exam and vital sign measurement, a new iPro® CGM device will be placed and will be worn for next 5 days. The subjects will maintain a diet history and will be given a One Touch glucometer and strips to check their blood glucose at home four times a day for next five days and log this onto the System Patient Log (included)

Subjects will undergo a MMTT, which includes consumption of a after a standard meal (Boost) + 5 grams of Glucomannan soluble fiber powder and scheduled blood draws over 3 hours.

For the next five days subjects will take 5 grams (1 teaspoon) of Glucomannan soluble fiber (provided by the investigator) three times a day with meals.

Visit 4: The subject will return to see the research coordinator for the CGM removal and data download from the device. At this time the study is completed.

ELIGIBILITY:
Inclusion Criteria:

1. Age: >18 year
2. Have undergone RNY Gastric Bypass >1 year.
3. Have symptoms of hypoglycemia (altered mental status or level of consciousness, with or without seizure, palpitations, tremor, anxiety/arousal, sweating, hunger, paresthesias, behavioral changes, fatigue, confusion), documented hypoglycemia (blood glucose<70 mg/dl), hypoglycemic unawareness (recurrent hypoglycemia without symptoms).

Exclusion Criteria:

1. Patient with Diabetes Type 1 or Type 2. Information identified during history taking or subject undergoing treatment of active diabetes.
2. Patient on medications or treatment (insulin, metformin, glyburide, diazoxide, octreotide, calcium channel blockers), which can cause hypoglycemia.
3. Patients with disorders, which can cause hypoglycemia, like untreated hypothyroidism, adrenal insufficiency, and growth hormone deficiency.
4. Complications of RNY i.e. Ulcers and hernia.
5. Current use of glucocorticoids or medications known to affect blood glucose levels.
6. Any patient that is unable to comply with dietary recommendations, technical iPro, glucometer actions or any part of the research protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: amy freeth, MD, Principal Investigator — Bassett Healthcare

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Baseline Phase (Control) and Treatment Phase (Glucomannan): Control:
  iPro® Continuous Glucose Monitor (CGM) device will be worn for 5 days. The subjects will maintain a diet history and will be given a One Touch glucometer and strips to check their blood glucose at home four times a day for next five days and log this onto the System Patient Log.
  Subjects will undergo Mixed Meal Tolerance Tests, which includes consumption of a standard meal (Boost) and scheduled blood draws over 3 hours.
  Glucomannan:
  iPro CGM device will be worn for 5 days. Subjects will maintain a diet history and will be given a One Touch glucometer and strips to check their blood glucose at home four times/day for next 5 days and log this onto the System Patient Log.
  Subjects will undergo Mixed Meal Tolerance Testing, which includes consumption of a standard meal (Boost) + 5 grams of Glucomannan soluble fiber powder and scheduled blood draws over 3 hours.
  glucomannan: Glucomannan is a natural, odorless soluble fiber that is found in the konjac plant.
Period: Overall Study
Arm/Group | Baseline Phase (Control) and Treatment Phase (Glucomannan)
Started | 11
Completed | 10
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Baseline Phase (Control), Crossover to Treatment (Glucomannan): Control:
  iPro CGM device will be worn for 5 days. The subjects will maintain a diet history and will be given a One Touch glucometer and strips to check their blood glucose at home four times a day for next five days and log this onto the System Patient Log.
  Glucomannan:
  For the next five days subjects will take the following amounts of Glucomannan soluble fiber (provided by the investigator) three times a day with meals.
  Breakfast: Take 5 grams (1 tsp) of Glucomannan. Lunch: Take 5 grams (1 tsp) of Glucomannan Dinner: Take 5 grams (1 tsp) of Glucomannan.
  glucomannan: Glucomannan is a natural, odorless soluble fiber that is found in the konjac plant.
Arm/Group | Baseline Phase (Control), Crossover to Treatment (Glucomannan)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Difference Score: Percent of Time Spent in Hypoglycemic State
Description: Percent of time within hypoglycemic blood glucose range (bg<70) compared between treatment (glucomannan) and control phases, as captured by the continuous glucose monitoring device. Difference score calculated as % time with bg<70 in treatment condition minus % time with bg<70 in control condition.
Time Frame: 10 days
Measure: Mean (Standard Deviation); unit: Difference score, trt-control (percent)
Groups:
- Baseline Phase (Control) and Treatment Phase (Glucomannan): Control:
  iPro CGM device will be worn for 5 days. The subjects will maintain a diet history and will be given a One Touch glucometer and strips to check their blood glucose at home four times a day for next five days and log this onto the System Patient Log.
  Subjects will undergo Mixed Meal Tolerance Tests, which includes consumption of a standard meal (Boost) and scheduled blood draws over 3 hours.
  Glucomannan:
  iPro CGM device will be worn for 5 days. Subjects will maintain a diet history and will be given a One Touch glucometer and strips to check their blood glucose at home four times/day for next 5 days and log this onto the System Patient Log.
  Subjects will undergo Mixed Meal Tolerance Testing, which includes consumption of a standard meal (Boost) + 5 grams of Glucomannan soluble fiber powder and scheduled blood draws over 3 hours.
  glucomannan: Glucomannan is a natural, odorless soluble fiber that is found in the konjac plant.
Arm/Group | Baseline Phase (Control) and Treatment Phase (Glucomannan)
Number analyzed (Participants) | 10
Difference score, trt-control (percent) | 1.2 (8.2)
Statistical Analysis 1: Comparison: Baseline Phase (Control) and Treatment Phase (Glucomannan); Test type: Superiority or Other; p = 0.99, Wilcoxon Signed Rank Test

2. Secondary Outcome: Difference Score: Percent of Time Within Normal Blood Glucose Limits
Description: Percent of time within normal blood glucose limits (bg 70-140) compared between treatment (glucomannan) and control phases, as captured by the continuous glucose monitoring device. Difference score calculated as % time within normal limits in treatment condition minus % time within normal limits in control condition.
Time Frame: 10 days
Measure: Mean (Standard Deviation); unit: Difference score, trt-control (percent)
Arm/Group | Baseline Phase (Control) and Treatment Phase (Glucomannan)
Number analyzed (Participants) | 10
Difference score, trt-control (percent) | -3.2 (7.5)
Statistical Analysis 1: Comparison: Baseline Phase (Control) and Treatment Phase (Glucomannan); Test type: Superiority or Other; p = 0.4922, Wilcoxon Signed Rank Test

3. Secondary Outcome: Difference Score: Percent of Time With Elevated Blood Glucose
Description: Percent of time within hyperglycemic blood glucose range (bg>140) compared between treatment (glucomannan) and control phases, as captured by the continuous glucose monitoring device. Difference score calculated as % time with bg>140 in treatment condition minus % time with bg>140 in control condition.
Time Frame: 10 days
Measure: Mean (Standard Deviation); unit: Difference score, trt-control (percent)
Arm/Group | Baseline Phase (Control) and Treatment Phase (Glucomannan)
Number analyzed (Participants) | 10
Difference score, trt-control (percent) | 2.0 (7.9)
Statistical Analysis 1: Comparison: Baseline Phase (Control) and Treatment Phase (Glucomannan); Test type: Superiority or Other; p = 0.77, Wilcoxon Signed Rank Test

4. Primary Outcome: Mixed Meal Testing: Difference Score: Blood Glucose Level (mg/dL)
Description: Difference score (trt-control) of blood glucose at 120 minutes post meal.
Time Frame: 120 minutes post-meal
Measure: Mean (Standard Deviation); unit: Difference score, trt-control (mg/dL)
Arm/Group | Baseline Phase (Control) and Treatment Phase (Glucomannan)
Number analyzed (Participants) | 8
Difference score, trt-control (mg/dL) | 5.25 (4.39)
Statistical Analysis 1: Comparison: Baseline Phase (Control) and Treatment Phase (Glucomannan); Test type: Superiority or Other; p = 0.0156, Wilcoxon Signed Rank Test

5. Primary Outcome: Mixed Meal Testing: Difference Score: Insulin Level (μU/mL)
Description: Difference score (trt-control) of insulin level at 30 minutes post meal.
Time Frame: 30 minutes post-meal
Measure: Mean (Standard Deviation); unit: Difference score, trt-control (μU/mL)
Arm/Group | Baseline Phase (Control) and Treatment Phase (Glucomannan)
Number analyzed (Participants) | 10
Difference score, trt-control (μU/mL) | -109.86 (79.47)
Statistical Analysis 1: Comparison: Baseline Phase (Control) and Treatment Phase (Glucomannan); Test type: Superiority or Other; p = 0.020, Wilcoxon Signed Rank Test

6. Primary Outcome: Mixed Meal Testing: Difference Score: Insulin Level (μU/mL)
Description: Difference score (trt-control) of insulin level at 60 minutes post meal.
Time Frame: 60 minutes post-meal
Measure: Mean (Standard Deviation); unit: Difference score, trt-control (μU/mL)
Arm/Group | Baseline Phase (Control) and Treatment Phase (Glucomannan)
Number analyzed (Participants) | 10
Difference score, trt-control (μU/mL) | -8.34 (13.41)
Statistical Analysis 1: Comparison: Baseline Phase (Control) and Treatment Phase (Glucomannan); Test type: Superiority or Other; p = 0.13, Wilcoxon Signed Rank Test

ADVERSE EVENTS:
Groups:
- Baseline Phase (Control) and Treatment Phase (Glucomannan): Control:
  iPro CGM device will be worn for 5 days. The subjects will maintain a diet history and will be given a One Touch glucometer and strips to check their blood glucose at home four times a day for next five days and log this onto the System Patient Log.
  Glucomannan:
  For the next five days subjects will take the following amounts of Glucomannan soluble fiber (provided by the investigator) three times a day with meals.
  Breakfast: Take 5 grams (1 tsp) of Glucomannan. Lunch: Take 5 grams (1 tsp) of Glucomannan Dinner: Take 5 grams (1 tsp) of Glucomannan.
  glucomannan: Glucomannan is a natural, odorless soluble fiber that is found in the konjac plant.
Arm/Group | Baseline Phase (Control) and Treatment Phase (Glucomannan)
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes